CLINICAL TRIAL: NCT00979589
Title: Randomized,Double-blind Trial Comparing the Effects of a 3-month Clopidogrel Regimen,Combined With ASA During the First 21days,Versus ASA Alone for the Acute Treatment of TIA or Minor Stroke
Brief Title: Clopidogrel in High-risk Patients With Acute Non-disabling Cerebrovascular Events
Acronym: CHANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008ZX09312-008
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: stroke; transient ischemic attack; acute treatment; acute non-disabling cerebrovascular event; clopidogrel; clopidogrel combined with ASA; recurrence of stroke and other vascular events
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Clopidogrel and asprin (Active Comparator)
  Interventions: Drug: Clopidogrel
- Asprin and placebo (Placebo Comparator)
  Interventions: Drug: Placebo of clopidogrel and Asprin

INTERVENTIONS:
Drug: Clopidogrel — The first group will receive a 300mg loading dose (LD) of clopidogrel on the day of randomization, followed by 75 mg clopidogrel/day from Day 2 to 3 months. ASA will be given in a total dose ranging between 75 mg and 300 mg (open label) on the first day, followed by blinded 75 mg once /day from Day 2 to Day 21st. Between Day 21st and 3-month visits, ASA 75 mg will be replaced by a placebo of ASA 75 mg.
  Other Names: Plavix
  Arms: Combination Clopidogrel and asprin
Drug: Placebo of clopidogrel and Asprin — The second group will receive open label ASA in a total dose ranging between 75 mg and 300 mg on the first day, followed by blinded 75 mg once /day from Day 2 to 3 months. A placebo for clopidogrel will be given from the day of randomization until the 3-month visit.
  Other Names: Acetylsalicylic acid
  Arms: Asprin and placebo

SUMMARY:
The purpose of this study is to assess the effects of a 3-month regimen of clopidogrel initiated with a loading dose (LD) of 300 mg followed by 75 mg/day during the first 21days versus a 3-month regimen of ASA 75 mg/day alone on reducing the 3-month risk of any stroke (both ischemic and hemorrhagic, primary outcome) when initiated within 24 hours of symptom onset in high-risk patients with TIA or minor stroke.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Adult subjects (male or female ≥ 40 years)
2. Acute non-disabling ischemic stroke (NIHSS≤3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle.
3. TIA (Neurological deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with study drug within 24 hours of symptoms onset and with moderate-to-high risk of stroke recurrence (ABCD2 score ≥ 4 at the time of randomization). Symptom onset is defined by the "last see normal" principle.
4. Informed consent signed

Primary Efficacy Endpoint:

Percentage of patients with the 3-month new vascular events, defined as any event of the following:Any stroke (ischemic or hemorrhage).

ELIGIBILITY:
Inclusion criteria:

* Adult subjects (male or female≥40 years)
* Acute non-disabling ischemic stroke (NIHSS≤3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* TIA (Neurological deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with study drug within 24 hours of symptoms onset and with moderate-to-high risk of stroke recurrence (ABCD2 score≥4 at the time of randomization).Symptom onset is defined by the "last see normal" principle
* Informed consent signed

Exclusion Criteria:

* Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head CT or MRI
* Isolated or pure sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI
* Modified Rankin Scale Score>2 at randomization (pre-morbid historical assessment)
* NIH Stroke Score≥4 at randomization
* Clear indication for anticoagulation(presumed cardiac source of embolus, e.g., atrial fibrillation, prosthetic cardiac valves known or suspected endocarditis)
* Contraindication to clopidogrel or ASA
* Known allergy
* Severe renal or hepatic insufficiency
* Severe cardiac failure, asthma
* Hemostatic disorder or systemic bleeding
* History of hemostatic disorder or systemic bleeding
* History of thrombocytopenia or neutropenia
* History of drug-induced hematologic or hepatic abnormalities
* Low white blood cell (<2 x109/l) or platelet count (<100 x109/l)
* Use of thrombolysis within 24 hours prior to randomization
* History of intracranial hemorrhage
* Anticipated requirement for long-term non-study antiplatelet drugs, or NSAIDs affecting platelet function
* Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anti coagulation
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months (if clinically indicated, vascular imaging should be performed prior to randomization whenever possible)
* Scheduled for surgery or interventional treatment requiring study drug cessation
* Qualifying TIA or minor stroke induced by angiography or surgery
* Severe non-cardiovascular comorbidity with life expectancy < 3 months
* Women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test
* Currently receiving an investigational drug or device

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5100 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with the 3-month new vascular events, defined as any event of the following: Any stroke (ischemic or hemorrhage) | 3 months

SECONDARY OUTCOMES:
Percentage of patients with the 3-month new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ MI/ vascular death) as a cluster and evaluated individually. | 3 months
Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6 at 3 month follow-up | 3 months
Further efficacy exploratory analysis:Impairment (changes in NIHSS scores at 3 month follow-up). | 3 months
Further efficacy exploratory analysis:Quality of Life (EuroQol EQ-5D scale) | 3 months
Efficacy endpoint will also be analyzed stratified by etiological subtypes, by time randomization (< 12 hours vs. ≥ 12 hours), by qualifying event (TIA vs. minor stroke), and by age | 3 months
Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage. | 3 months
Incidence symptomatic and asymptomatic intracranial hemorrhagic events at 3 months | 3 months
Intracranial hemorrhage | 3 months
Total mortality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun NA Wang, M.D, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China; S.Claiborne NA Johnston, M.D, Ph.D, Principal Investigator — Departments of Neurology, Epidemiology, University of California, San Francisco, USA
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Wang Y, Johnston SC; CHANCE Investigators. Rationale and design of a randomized, double-blind trial comparing the effects of a 3-month clopidogrel-aspirin regimen versus aspirin alone for the treatment of high-risk patients with acute nondisabling cerebrovascular event. Am Heart J. 2010 Sep;160(3):380-386.e1. doi: 10.1016/j.ahj.2010.05.017. PMID 20826243
- [Background] Wang Y, Zhao X, Lin J, Li H, Johnston SC, Lin Y, Pan Y, Liu L, Wang D, Wang C, Meng X, Xu J, Wang Y; CHANCE investigators. Association Between CYP2C19 Loss-of-Function Allele Status and Efficacy of Clopidogrel for Risk Reduction Among Patients With Minor Stroke or Transient Ischemic Attack. JAMA. 2016 Jul 5;316(1):70-8. doi: 10.1001/jama.2016.8662. PMID 27348249
- [Background] Jing J, Meng X, Zhao X, Liu L, Wang A, Pan Y, Li H, Wang D, Johnston SC, Wang Y, Wang Y. Dual Antiplatelet Therapy in Transient Ischemic Attack and Minor Stroke With Different Infarction Patterns: Subgroup Analysis of the CHANCE Randomized Clinical Trial. JAMA Neurol. 2018 Jun 1;75(6):711-719. doi: 10.1001/jamaneurol.2018.0247. PMID 29582084
- [Background] Pan Y, Elm JJ, Li H, Easton JD, Wang Y, Farrant M, Meng X, Kim AS, Zhao X, Meurer WJ, Liu L, Dietrich D, Wang Y, Johnston SC. Outcomes Associated With Clopidogrel-Aspirin Use in Minor Stroke or Transient Ischemic Attack: A Pooled Analysis of Clopidogrel in High-Risk Patients With Acute Non-Disabling Cerebrovascular Events (CHANCE) and Platelet-Oriented Inhibition in New TIA and Minor Ischemic Stroke (POINT) Trials. JAMA Neurol. 2019 Dec 1;76(12):1466-1473. doi: 10.1001/jamaneurol.2019.2531. PMID 31424481
- [Background] Pan Y, Meng X, Jing J, Li H, Zhao X, Liu L, Wang D, Johnston SC, Wang Y, Wang Y; CHANCE Investigators. Association of multiple infarctions and ICAS with outcomes of minor stroke and TIA. Neurology. 2017 Mar 14;88(11):1081-1088. doi: 10.1212/WNL.0000000000003719. Epub 2017 Feb 15. PMID 28202699
- [Background] Pan Y, Jing J, Chen W, Meng X, Li H, Zhao X, Liu L, Wang D, Johnston SC, Wang Y, Wang Y; CHANCE investigators. Risks and benefits of clopidogrel-aspirin in minor stroke or TIA: Time course analysis of CHANCE. Neurology. 2017 May 16;88(20):1906-1911. doi: 10.1212/WNL.0000000000003941. Epub 2017 Apr 19. PMID 28424269
- [Background] Li J, Wang A, Zhao X, Liu L, Meng X, Lin J, Jing J, Zou X, Wang Y, Wang Y; CHANCE Investigators. High-sensitive C-reactive protein and dual antiplatelet in intracranial arterial stenosis. Neurology. 2018 Feb 6;90(6):e447-e454. doi: 10.1212/WNL.0000000000004928. Epub 2018 Jan 12. PMID 29330312
- [Result] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Derived] Han C, Yang M, Pan Y, Li H, Liu L, Meng X, Wang Y, Wang Y. Disabling Neurologic Deficits and Antiplatelet Therapy in Acute Minor Stroke. J Am Heart Assoc. 2025 Apr 15;14(8):e029734. doi: 10.1161/JAHA.122.029734. Epub 2025 Apr 7. PMID 40194961
- [Derived] Qiu X, Jiang Y, Gu HQ, Jiang Y, Huang X, Meng X, Wang Y, Li Z. Polygenic Risk Score for the Efficacy of Clopidogrel in Patients With Minor Stroke or Transient Ischemic Attack: A Post Hoc Analysis of the CHANCE Trial. Stroke. 2025 Apr;56(4):818-827. doi: 10.1161/STROKEAHA.124.049140. Epub 2025 Mar 7. PMID 40052280
- [Derived] Yang M, Xu J, Xue J, Pan Y, Cheng A, Gao F, Meng X, Miao Z, Wang Y, Wang Y; CHANCE Investigators. Efficacy of dual antiplatelet therapy after ischemic stroke according to hsCRP levels and CYP2C19 genotype. Am Heart J. 2025 Feb;280:89-97. doi: 10.1016/j.ahj.2024.10.017. Epub 2024 Nov 12. PMID 39536847
- [Derived] Qiu X, Zhang Y, Gu H, Jiang Y, Pan Y, Jiang Y, Meng X, Wang Y, Zhao X, Li H, Wang X, Wang Y, Li Z; CHANCE Investigators. Association Between CYP2B6 Polymorphisms and Efficacy of Clopidogrel in Minor Stroke or Transient Ischemic Attack. Stroke. 2023 Jul;54(7):1770-1776. doi: 10.1161/STROKEAHA.122.040507. Epub 2023 Jun 2. PMID 37264909
- [Derived] Chen P, Wu Q, Xie X, Jing J, Gu H, Wang X, Meng X, Liu L, Wang Y, Wang Y; CHANCE Investigators. Systolic blood pressure and recurrent stroke in patients with different lesion patterns on diffusion weighted imaging. J Clin Hypertens (Greenwich). 2022 Oct;24(10):1350-1357. doi: 10.1111/jch.14543. Epub 2022 Aug 12. PMID 35959564
- [Derived] Zhang X, Jing J, Zhao X, Liu L, Wang A, Pan Y, Wang D, Johnston SC, Wang Y, Wang Y, Meng X. No rebound effect after a course of clopidogrel in patients with acute TIA or minor stroke. Neurol Res. 2022 Nov;44(11):957-963. doi: 10.1080/01616412.2022.2075660. Epub 2022 Jun 13. PMID 35695332
- [Derived] Pan Y, Wangqin R, Li H, Jin A, Li J, Lin J, Meng X, Xian Y, Laskowitz DT, Wang Y. LDL-C levels, lipid-lowering treatment and recurrent stroke in minor ischaemic stroke or TIA. Stroke Vasc Neurol. 2022 Aug;7(4):276-284. doi: 10.1136/svn-2021-001317. Epub 2022 Mar 7. PMID 35256525
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Pan Y, Wangqin R, Li H, Wang Y, Meng X, Johnston SC, Simon T, Lin J, Zhao X, Liu L, Wang D, Wang Y. F2R Polymorphisms and Clopidogrel Efficacy and Safety in Patients With Minor Stroke or TIA. Neurology. 2021 Jan 5;96(1):e1-e9. doi: 10.1212/WNL.0000000000011078. Epub 2020 Oct 22. PMID 33093222
- [Derived] Wang G, Jing J, Li J, Pan Y, Yan H, Meng X, Zhao X, Liu L, Li H, Wang DZ, Wang Y, Wang Y. Association of elevated hs-CRP and multiple infarctions with outcomes of minor stroke or TIA: subgroup analysis of CHANCE randomised clinical trial. Stroke Vasc Neurol. 2021 Mar;6(1):80-86. doi: 10.1136/svn-2020-000369. Epub 2020 Sep 21. PMID 32958697
- [Derived] Chen H, Pan Y, Zong L, Jing J, Meng X, Xu Y, Yan H, Zhao X, Liu L, Li H, Johnston SC, Wang Y, Wang Y. Cerebral small vessel disease or intracranial large vessel atherosclerosis may carry different risk for future strokes. Stroke Vasc Neurol. 2020 Jun;5(2):128-137. doi: 10.1136/svn-2019-000305. Epub 2020 Apr 15. PMID 32606085
- [Derived] Xu YY, Zong LX, Zhang CQ, Pan YS, Jing J, Meng X, Li H, Zhao XQ, Liu LP, Wang D, Wang YL, Wang YJ; CHANCE Investigators. The association of white matter hyperintensities with stroke outcomes and antiplatelet therapy in minor stroke patients. Ann Transl Med. 2020 Mar;8(6):331. doi: 10.21037/atm.2020.02.137. PMID 32355775
- [Derived] Li J, Wang Y, Li H, Zuo Z, Lin J, Wang A, Zhao X, Liu L, Wang Y; CHANCE Investigators. Homocysteine Level Predicts Response to Dual Antiplatelet in Women With Minor Stroke or Transient Ischemic Attack: Subanalysis of the CHANCE Trial. Arterioscler Thromb Vasc Biol. 2020 Mar;40(3):839-846. doi: 10.1161/ATVBAHA.119.313741. Epub 2020 Jan 16. PMID 31941381
- [Derived] Yang M, Wang A, Li J, Zhao X, Liu L, Meng X, Jing J, Zhang N, Johnston SC, Wang Y, Wang Y. Lp-PLA2 and dual antiplatelet agents in intracranial arterial stenosis. Neurology. 2020 Jan 14;94(2):e181-e189. doi: 10.1212/WNL.0000000000008733. Epub 2019 Dec 10. PMID 31822574
- [Derived] Mo J, Chen Z, Xu J, Wang A, Dai L, Cheng A, Meng X, Li H, Wang Y; CHANCE Investigators. Efficacy of Clopidogrel-Aspirin Therapy for Stroke Does Not Exist in CYP2C19 Loss-of-Function Allele Noncarriers With Overweight/Obesity. Stroke. 2020 Jan;51(1):224-231. doi: 10.1161/STROKEAHA.119.026845. Epub 2019 Nov 15. PMID 31726963
- [Derived] Chen W, Pan Y, Jing J, Zhao X, Liu L, Meng X, Wang Y, Lin Y, Wang Y; CHANCE Investigators. Association of Body Mass Index and Risk of Stroke After Acute Minor Stroke or TIA: a Post Hoc Analysis of a Randomized Controlled Trial. Neurotox Res. 2019 Nov;36(4):836-843. doi: 10.1007/s12640-019-00056-4. Epub 2019 May 24. PMID 31127478
- [Derived] Xie X, Wang X, Laskowitz DT, Zhao X, Miao Z, Liu L, Li H, Meng X, Wang Y, Wang Y; CHANCE investigators. Effect of dual versus mono antiplatelet therapy on recurrent stroke modulated by activated partial thromboplastin time. Eur J Neurol. 2019 Sep;26(9):1168-e78. doi: 10.1111/ene.13961. Epub 2019 May 9. PMID 30972875
- [Derived] Pan Y, Chen W, Wang Y, Li H, Johnston SC, Simon T, Zhao X, Liu L, Wang D, Meng X, Wang Y; Clopidogrel in High-Risk Patients With Acute Nondisabling Cerebrovascular Events (CHANCE) Investigators. Association Between ABCB1 Polymorphisms and Outcomes of Clopidogrel Treatment in Patients With Minor Stroke or Transient Ischemic Attack: Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2019 May 1;76(5):552-560. doi: 10.1001/jamaneurol.2018.4775. PMID 30742211
- [Derived] Wang G, Jing J, Pan Y, Meng X, Zhao X, Liu L, Li H, Wang D, Wang Y, Wang Y; CHANCE Investigatores. Does all single infarction have lower risk of stroke recurrence than multiple infarctions in minor stroke? BMC Neurol. 2019 Jan 8;19(1):7. doi: 10.1186/s12883-018-1215-0. PMID 30621613
- [Derived] Wang A, Li S, Zhang N, Dai L, Zuo Y, Wang Y, Meng X, Wang Y. Oxidized Low-Density Lipoprotein to High-Density Lipoprotein Ratio Predicts Recurrent Stroke in Minor Stroke or Transient Ischemic Attack. Stroke. 2018 Nov;49(11):2637-2642. doi: 10.1161/STROKEAHA.118.022077. PMID 30355199
- [Derived] Zhu B, Liu H, Pan Y, Jing J, Li H, Zhao X, Liu L, Wang D, Johnston SC, Wang Z, Wang Y, Wang Y; CHANCE Investigators. Elevated Neutrophil and Presence of Intracranial Artery Stenosis Increase the Risk of Recurrent Stroke. Stroke. 2018 Oct;49(10):2294-2300. doi: 10.1161/STROKEAHA.118.022126. PMID 30355101
- [Derived] Wang A, Xu J, Chen G, Wang D, Johnston SC, Meng X, Lin J, Li H, Cao Y, Zhang N, Ma C, Dai L, Zhao X, Liu L, Wang Y, Wang Y. Oxidized low-density lipoprotein predicts recurrent stroke in patients with minor stroke or TIA. Neurology. 2018 Sep 4;91(10):e947-e955. doi: 10.1212/WNL.0000000000006118. Epub 2018 Aug 8. PMID 30089614
- [Derived] Ma Y, Liu Y, Xu J, Wang Y, Wang Y, Du F. Effect of dual antiplatelet on recurrent stroke in minor stroke or TIA depends on bodyweight. Ther Clin Risk Manag. 2018 May 8;14:861-870. doi: 10.2147/TCRM.S156694. eCollection 2018. PMID 29773949
- [Derived] Wangqin R, Wang X, Wang Y, Xian Y, Zhao X, Liu L, Li H, Meng X, Wang Y. Risk factors associated with 90-day recurrent stroke in patients on dual antiplatelet therapy for minor stroke or high-risk TIA: a subgroup analysis of the CHANCE trial. Stroke Vasc Neurol. 2017 Jul 6;2(4):176-183. doi: 10.1136/svn-2017-000088. eCollection 2017 Dec. PMID 29507777
- [Derived] Pan Y, Cai X, Jing J, Meng X, Li H, Wang Y, Zhao X, Liu L, Wang D, Johnston SC, Wei T, Wang Y; CHANCE Investigators. Stress Hyperglycemia and Prognosis of Minor Ischemic Stroke and Transient Ischemic Attack: The CHANCE Study (Clopidogrel in High-Risk Patients With Acute Nondisabling Cerebrovascular Events). Stroke. 2017 Nov;48(11):3006-3011. doi: 10.1161/STROKEAHA.117.019081. PMID 29051218
- [Derived] Wang D, Gui L, Dong Y, Li H, Li S, Zheng H, Wang A, Meng X, Liu LP, Wang YL, Wang G, Jing J, Li Z, Zhao XQ, Wang YJ. Dual antiplatelet therapy may increase the risk of non-intracranial haemorrhage in patients with minor strokes: a subgroup analysis of the CHANCE trial. Stroke Vasc Neurol. 2016 Jun 24;1(2):29-36. doi: 10.1136/svn-2016-000008. eCollection 2016 Jun. PMID 28959461
- [Derived] Lin Y, Wang A, Li J, Lin J, Wang D, Meng X, Ou L, Chen W, Zhao X, Liu L, Wang Y, Wang Y; CHANCE Investigators. Impact of Glycemic Control on Efficacy of Clopidogrel in Transient Ischemic Attack or Minor Stroke Patients With CYP2C19 Genetic Variants. Stroke. 2017 Apr;48(4):998-1004. doi: 10.1161/STROKEAHA.116.016463. Epub 2017 Mar 13. PMID 28289237
- [Derived] Zhou Y, Pan Y, Wu Y, Zhao X, Li H, Wang D, Johnston SC, Liu L, Wang C, Meng X, Wang Y, Wang Y; CHANCE Investigators. Effect of Estimated Glomerular Filtration Rate Decline on the Efficacy and Safety of Clopidogrel With Aspirin in Minor Stroke or Transient Ischemic Attack: CHANCE Substudy (Clopidogrel in High-Risk Patients With Acute Nondisabling Cerebrovascular Events). Stroke. 2016 Nov;47(11):2791-2796. doi: 10.1161/STROKEAHA.116.014761. Epub 2016 Oct 13. PMID 27738237
- [Derived] Pan Y, Jing J, Li H, Wang Y, Wang Y, He Y; CHANCE investigators. Abnormal glucose regulation increases stroke risk in minor ischemic stroke or TIA. Neurology. 2016 Oct 11;87(15):1551-1556. doi: 10.1212/WNL.0000000000003200. Epub 2016 Sep 9. PMID 27613582
- [Derived] Li J, Zhao X, Meng X, Lin J, Liu L, Wang C, Wang A, Wang Y, Wang Y; CHANCE Investigators. High-Sensitive C-Reactive Protein Predicts Recurrent Stroke and Poor Functional Outcome: Subanalysis of the Clopidogrel in High-Risk Patients With Acute Nondisabling Cerebrovascular Events Trial. Stroke. 2016 Aug;47(8):2025-30. doi: 10.1161/STROKEAHA.116.012901. Epub 2016 Jun 21. PMID 27328699
- [Derived] Li Z, Wang Y, Zhao X, Liu L, Wang D, Wang C, Meng X, Li H, Pan Y, Wang X, Wang C, Yang X, Zhang C, Jing J, Xian Y, Johnston SC, Wang Y; CHANCE Investigators. Treatment Effect of Clopidogrel Plus Aspirin Within 12 Hours of Acute Minor Stroke or Transient Ischemic Attack. J Am Heart Assoc. 2016 Mar 21;5(3):e003038. doi: 10.1161/JAHA.115.003038. PMID 27001965
- [Derived] Liu L, Wong KS, Leng X, Pu Y, Wang Y, Jing J, Zou X, Pan Y, Wang A, Meng X, Wang C, Zhao X, Soo Y, Johnston SC, Wang Y; CHANCE Investigators. Dual antiplatelet therapy in stroke and ICAS: Subgroup analysis of CHANCE. Neurology. 2015 Sep 29;85(13):1154-62. doi: 10.1212/WNL.0000000000001972. PMID 26330567
- [Derived] Li J, Wang Y, Lin J, Wang D, Wang A, Zhao X, Liu L, Wang C, Wang Y; CHANCE Investigators. Soluble CD40L Is a Useful Marker to Predict Future Strokes in Patients With Minor Stroke and Transient Ischemic Attack. Stroke. 2015 Jul;46(7):1990-2. doi: 10.1161/STROKEAHA.115.008685. Epub 2015 May 26. PMID 26012640
- [Derived] Wang Y, Pan Y, Zhao X, Li H, Wang D, Johnston SC, Liu L, Meng X, Wang A, Wang C, Wang Y; CHANCE Investigators. Clopidogrel With Aspirin in Acute Minor Stroke or Transient Ischemic Attack (CHANCE) Trial: One-Year Outcomes. Circulation. 2015 Jul 7;132(1):40-6. doi: 10.1161/CIRCULATIONAHA.114.014791. Epub 2015 May 8. PMID 25957224